CLINICAL TRIAL: NCT01252186
Title: A Multinational, Multicenter, Randomized, Open-Label Study to Evaluate the Impact of a 91-Day Extended Cycle Oral Contraceptive Regimen, Compared to Two 28-day Standard Oral Contraceptive Regimens, on Hemostatic Parameters in Healthy Women.
Brief Title: A Multicenter Study to Evaluate the Effects of a 91-Day Extended Cycle Oral Contraceptive on Hemostatic Parameters in Healthy Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Teva Women's Health (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PSE-HSP-203; 2010-023215-34 (EudraCT Number)
Record Dates: First submitted 2010-11-30; First posted 2010-12-02 (Estimated); Results first posted 2015-03-13 (Estimated); Last update posted 2015-03-13 (Estimated); Status verified 2015-02

CONDITIONS: Hemostasis; Oral Contraceptive
Keywords: Contraception; Hemostasis; Blood Coagulation
MeSH Terms: conditions — Thrombosis | interventions — Seasonique; Desogestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 91-day Levonorgestrel Oral Contraceptive (Experimental): Participants received 12 weeks (84 consecutive days) of active combination tablets containing 150 µg levonorgestrel (LNG)/30 µg ethinyl estradiol (EE), followed by 7 days of 10 µg EE monotherapy in each 91-day cycle for a total of two 91-day cycles.
  Interventions: Drug: 91-day Levonorgestrel Oral Contraceptive
- 28-day Levonorgestrel Oral Contraceptive (Active Comparator): Participants received 21 days of active combination tablets containing 150 µg LNG/30 µg EE, followed by no treatment for 7 days in each 28-day cycle for a total of six 28-day cycles.
  Interventions: Drug: 28-day Levonorgestrel Oral Contraceptive
- 28-day Desogestrel Oral Contraceptive (Active Comparator): Participants received 21 days of active combination tablets (containing 150 µg desogestrel (DSG)/30 µg EE, followed by no treatment for 7 days in each 28-day cycle for a total of six 28-day cycles.
  Interventions: Drug: 28-day Desogestrel Oral Contraceptive

INTERVENTIONS:
Drug: 91-day Levonorgestrel Oral Contraceptive — 91-day treatment consisting of 84 blue combination tablets containing 150 µg LNG/30 µg EE and 7 yellow tablets containing 10 µg EE.
  Other Names: Seasonique®
  Arms: 91-day Levonorgestrel Oral Contraceptive
Drug: 28-day Levonorgestrel Oral Contraceptive — 21 combination tablets containing 150 µg LNG/30 µg EE.
  Other Names: Minidril®
  Arms: 28-day Levonorgestrel Oral Contraceptive
Drug: 28-day Desogestrel Oral Contraceptive — 21 combination tablets containing 150 µg DSG/30 µg EE.
  Other Names: Marvelon®
  Arms: 28-day Desogestrel Oral Contraceptive

SUMMARY:
This study is being conducted to evaluate the impact of a 91-day extended cycle oral contraceptive compared to two 28-day oral contraceptive regimens on hemostatic parameters in healthy women.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal, non-pregnant, non-lactating women age 18-40 years old
* Body Mass Index (BMI) ≥18 kg/m² and <30 kg/m²
* Regular spontaneous menstrual cycle
* Others as dictated by FDA-approved protocol

Exclusion Criteria:

* Any condition which contraindicates the use of combination oral contraceptives
* Any history of, or active, deep vein thrombosis, pulmonary embolism, or arterial thromboembolic disease within one year of screening
* Any known genetic component for thrombophilia including Factor V Leiden mutation, prothrombin mutation, protein C deficiency, protein S deficience, or antithrombin III deficiency
* Others as dictated by FDA-approved protocol

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 265 (Actual)
Dates: Start 2010-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Women's Health Research Protocol Chair, Study Chair — Teva Women's Health Research
Locations (22):
- United States (19):
  - Teva Investigational Site, San Diego, California
  - Teva Investigational Site, Washington D.C., District of Columbia
  - Teva Investigational Site, Miami, Florida
  - Teva Investigational Site, West Palm Beach, Florida
  - Teva Investigational Site, Sandy Springs, Georgia
  - Teva Investigational Site, Edison, New Jersey
  - Teva Investigational Site, Plainsboro, New Jersey
  - Teva Investigational Site, Albuquerque, New Mexico
  - Teva Investigational Site, Port Jefferson, New York
  - Teva Investigational Site, Rochester, New York
  - Teva Investigational Site, Winston-Salem, North Carolina
  - Teva Investigational Site, Philadelphia, Pennsylvania
  - Teva Investigational Site, Pittsburgh, Pennsylvania
  - Teva Investigational Site, Uniontown, Pennsylvania
  - Teva Investigational Site, Dallas, Texas
  - Teva Investigational Site, Houston, Texas
  - Teva Investigational Site, San Antonio, Texas
  - Teva Investigational Site, Richmond, Virginia
  - Teva Investigational Site, Seattle, Washington
- Italy (3):
  - Teva Investigational Site, Cagliari
  - Teva Investigational Site, Modena
  - Teva Investigational Site, Pavia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 91-day Levonorgestrel Oral Contraceptive | 28-day Levonorgestrel Oral Contraceptive | 28-day Desogestrel Oral Contraceptive
Started | 87 | 91 | 87
Received Study Drug | 83 | 89 | 80
Completed | 57 | 59 | 53
Not Completed | 30 | 32 | 34
Not completed — Adverse Event | 9 | 6 | 8
Not completed — Withdrawal by Subject | 2 | 5 | 2
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Non-compliance | 0 | 3 | 4
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Pregnancy | 2 | 2 | 0
Not completed — Sponsor Request | 2 | 1 | 0
Not completed — Lost to Follow-up | 10 | 10 | 11
Not completed — Other - Miscellaneous Reasons | 5 | 5 | 7

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population included all randomized and treated participants who had both baseline and at least one post-baseline measurement of prothrombin fragment 1+2 (F1+2).
Groups:
- Total: Total of all reporting groups
Arm/Group | 91-day Levonorgestrel Oral Contraceptive | 28-day Levonorgestrel Oral Contraceptive | 28-day Desogestrel Oral Contraceptive | Total
Number analyzed (Participants) | 75 | 80 | 71 | 226
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.3 (5.87) | 26.8 (6.22) | 27.0 (5.75) | 27.0 (5.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 80 | 71 | 226
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1 | 5 | 3 | 9
  Black or African-American | 18 | 15 | 9 | 42
  Caucasian | 42 | 39 | 40 | 121
  Hispanic | 13 | 20 | 19 | 52
  Other | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to End of Month 6 in Prothrombin Fragment 1+2 Levels
Description: Prothrombin fragment 1+2 is a coagulation factor, released when prothrombin is cleaved by activated factor X. Elevated plasma levels of prothrombin fragment 1+2 indicate high risk of thrombosis.
Time Frame: Baseline to Month 6
Population: Per-Protocol (PP) Population included all data from ITT participants obtained prior to experiencing major protocol violations.
Measure: Least Squares Mean (Standard Error); unit: pmol/L
Arm/Group | 91-day Levonorgestrel Oral Contraceptive | 28-day Levonorgestrel Oral Contraceptive | 28-day Desogestrel Oral Contraceptive
Number analyzed (Participants) | 61 | 67 | 59
pmol/L | 169.53 (155.15) | 157.99 (150.11) | 592.29 (160.32)
Statistical Analysis 1: Comparison: 91-day Levonorgestrel Oral Contraceptive vs 28-day Levonorgestrel Oral Contraceptive; The primary endpoint was analyzed using a maximum likelihood-based mixed model repeated measures (MMRM) analysis of covariance (ANCOVA) with covariate adjustment for baseline, treatment, month, and the treatment-by-month interaction; Test type: Non-Inferiority or Equivalence — A conclusion of non-inferiority was reached if the lower limit of the confidence interval for the comparison (active control minus 91-day Levonorgestrel) was greater than -0.13 nmol/L (130 pmol/L); p = 0.958, Mixed Models Analysis; Treatment Difference = -11.54, 95% CI 2-sided [-440.1 to 417.0] — Treatment difference is calculated as (28-day Levonorgestrel - 91-day Levonorgestrel)
Statistical Analysis 2: Comparison: 91-day Levonorgestrel Oral Contraceptive vs 28-day Desogestrel Oral Contraceptive; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.060, Mixed Models Analysis; Treatment Difference = 422.76, 95% CI 2-sided [-18.3 to 863.8] — Treatment difference is calculated as (28-day Desogestrel - 91-day Levonorgestrel)

2. Secondary Outcome: Change From Baseline to End of Month 6 in D-dimer
Description: D-dimer is the degradation product of cross-linked fibrin and is a marker of thrombin and fibrin formation and turnover.
Time Frame: Baseline to Month 6
Population: Per-protocol population
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | 91-day Levonorgestrel Oral Contraceptive | 28-day Levonorgestrel Oral Contraceptive | 28-day Desogestrel Oral Contraceptive
Number analyzed (Participants) | 61 | 67 | 59
ng/mL | 86.74 (31.49) | 72.43 (30.18) | 158.05 (32.07)
Statistical Analysis 1: Comparison: 91-day Levonorgestrel Oral Contraceptive vs 28-day Levonorgestrel Oral Contraceptive; The endpoint was analyzed using a maximum likelihood-based mixed model repeated measures (MMRM) analysis of covariance (ANCOVA) with covariate adjustment for baseline, treatment, month, and the treatment-by-month interaction; Test type: Superiority or Other; p = 0.745, Mixed Models Analysis; Treatment Difference = -14.31, 95% CI 2-sided [-100.8 to 72.2] — Treatment difference is calculated as (28-day Levonorgestrel - 91-day Levonorgestrel)
Statistical Analysis 2: Comparison: 91-day Levonorgestrel Oral Contraceptive vs 28-day Desogestrel Oral Contraceptive; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.115, Mixed Models Analysis; Treatment Difference = 71.31, 95% CI 2-sided [-17.5 to 160.1] — Treatment difference is calculated as (28-day Desogestrel - 91-day Levonorgestrel)

3. Secondary Outcome: Change From Baseline to End of Month 6 in Plasmin-Antiplasmin (PAP) Complex
Description: The plasmin-antiplasmin (PAP) complex is a marker of thrombin and fibrin formation and turnover.
Time Frame: Baseline to Month 6
Population: Per-protocol population
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | 91-day Levonorgestrel Oral Contraceptive | 28-day Levonorgestrel Oral Contraceptive | 28-day Desogestrel Oral Contraceptive
Number analyzed (Participants) | 61 | 67 | 59
ng/mL | 10.72 (44.55) | -6.42 (43.11) | 107.81 (45.97)
Statistical Analysis 1: Comparison: 91-day Levonorgestrel Oral Contraceptive vs 28-day Levonorgestrel Oral Contraceptive; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.782, Mixed Models Analysis; Treatment Difference = -17.14, 95% CI 2-sided [-139.4 to 105.1] — Treatment difference is calculated as (28-day Levonorgestrel - 91-day Levonorgestrel)
Statistical Analysis 2: Comparison: 91-day Levonorgestrel Oral Contraceptive vs 28-day Desogestrel Oral Contraceptive; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.131, Mixed Models Analysis; Treatment Difference = 97.09, 95% CI 2-sided [-29.2 to 223.4] — Treatment difference is calculated as (28-day Desogestrel - 91-day Levonorgestrel)

4. Secondary Outcome: Change From Baseline to End of Month 6 in Activated Partial Thromboplastin Time (APTT) Based Activated Protein-C Resistance (APC)
Description: The APC resistance assay is a clotting test that measures the ratio of APTT clotting times in the presence and absence of a standard amount of exogenous APC. APC resistance is calculated as the ratio of the clotting time after APC addition over the clotting time with no APC addition.
  APC resistance is defined as a poor anticoagulant response of plasma to APC (minimal prolongation of the APTT) and a correspondingly low ratio.
Time Frame: Baseline to Month 6
Population: Per-protocol population with available data
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | 91-day Levonorgestrel Oral Contraceptive | 28-day Levonorgestrel Oral Contraceptive | 28-day Desogestrel Oral Contraceptive
Number analyzed (Participants) | 61 | 67 | 58
ratio | -0.12 (0.04) | -0.15 (0.03) | -0.27 (0.04)
Statistical Analysis 1: Comparison: 91-day Levonorgestrel Oral Contraceptive vs 28-day Levonorgestrel Oral Contraceptive; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.428, Mixed Models Analysis; Treatment Difference = -0.04, 95% CI 2-sided [-0.1 to 0.1] — Treatment difference is calculated as (28-day Levonorgestrel - 91-day Levonorgestrel)
Statistical Analysis 2: Comparison: 91-day Levonorgestrel Oral Contraceptive vs 28-day Desogestrel Oral Contraceptive; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis; Treatment Difference = -0.16, 95% CI 2-sided [-0.3 to -0.1] — Treatment difference is calculated as (28-day Desogestrel - 91-day Levonorgestrel)

5. Secondary Outcome: Change From Baseline to End of Month 6 in Endogenous Thrombin Potential (EPT) Based Activated Protein-C Resistance (APC)
Description: This assay is based on measurement of the effect of activated protein C on the endogenous thrombin potential, the time integral of thrombin generation initiated in plasma through the extrinsic coagulation pathway.
  The APC resistance assay measures the ratio of endogenous thrombin potential in the presence and absence of a standard amount of exogenous APC.
  APC resistance is calculated as the ratio of EPT after APC addition over the EPT with no APC addition.
  APC resistance is defined as a poor anticoagulant response of plasma to APC (less inhibition of thrombin formation) and a correspondingly higher ratio.
Time Frame: Baseline to Month 6
Population: Per-protocol population
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | 91-day Levonorgestrel Oral Contraceptive | 28-day Levonorgestrel Oral Contraceptive | 28-day Desogestrel Oral Contraceptive
Number analyzed (Participants) | 61 | 67 | 59
ratio | 0.38 (0.05) | 0.37 (0.05) | 0.57 (0.05)
Statistical Analysis 1: Comparison: 91-day Levonorgestrel Oral Contraceptive vs 28-day Levonorgestrel Oral Contraceptive; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.868, Mixed Models Analysis; Treatment Difference = -0.01, 95% CI 2-sided [-0.2 to 0.1] — Treatment difference is calculated as (28-day Levonorgestrel - 91-day Levonorgestrel)
Statistical Analysis 2: Comparison: 91-day Levonorgestrel Oral Contraceptive vs 28-day Desogestrel Oral Contraceptive; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.012, Mixed Models Analysis; Treatment Difference = 0.20, 95% CI 2-sided [0.0 to 0.3] — Treatment difference is calculated as (28-day Desogestrel - 91-day Levonorgestrel)

6. Secondary Outcome: Change From Baseline to End of Month 6 in Fibrinogen
Description: Fibrinogen (factor I) is a glycoprotein that helps in the formation of blood clots.
Time Frame: Baseline to Month 6
Population: Per-protocol population
Measure: Least Squares Mean (Standard Error); unit: g/L
Arm/Group | 91-day Levonorgestrel Oral Contraceptive | 28-day Levonorgestrel Oral Contraceptive | 28-day Desogestrel Oral Contraceptive
Number analyzed (Participants) | 61 | 67 | 59
g/L | 0.12 (0.07) | 0.22 (0.06) | -0.04 (0.07)
Statistical Analysis 1: Comparison: 91-day Levonorgestrel Oral Contraceptive vs 28-day Levonorgestrel Oral Contraceptive; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.317, Mixed Models Analysis; Treatment Difference = 0.09, 95% CI 2-sided [-0.1 to 0.3] — Treatment difference is calculated as (28-day Levonorgestrel - 91-day Levonorgestrel)
Statistical Analysis 2: Comparison: 91-day Levonorgestrel Oral Contraceptive vs 28-day Desogestrel Oral Contraceptive; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.081, Mixed Models Analysis; Treatment Difference = -0.16, 95% CI 2-sided [-0.4 to 0.0] — Treatment difference is calculated as (28-day Desogestrel - 91-day Levonorgestrel)

7. Secondary Outcome: Change From Baseline to End of Month 6 in Plasminogen
Description: Plasminogen is the precursor of plasmin, which lyses fibrin clots.
Time Frame: Baseline to Month 6
Population: Per-protocol population
Measure: Least Squares Mean (Standard Error); unit: g/L
Arm/Group | 91-day Levonorgestrel Oral Contraceptive | 28-day Levonorgestrel Oral Contraceptive | 28-day Desogestrel Oral Contraceptive
Number analyzed (Participants) | 61 | 67 | 59
g/L | 0.04 (0.00) | 0.04 (0.00) | 0.04 (0.00)
Statistical Analysis 1: Comparison: 91-day Levonorgestrel Oral Contraceptive vs 28-day Levonorgestrel Oral Contraceptive; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.331, Mixed Models Analysis; Treatment Difference = -0.004, 95% CI 2-sided [-0.013 to 0.004] — Treatment difference is calculated as (28-day Levonorgestrel - 91-day Levonorgestrel)
Statistical Analysis 2: Comparison: 91-day Levonorgestrel Oral Contraceptive vs 28-day Desogestrel Oral Contraceptive; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.173, Mixed Models Analysis; Treatment Difference = -0.006, 95% CI 2-sided [-0.015 to 0.003] — Treatment difference is calculated as (28-day Desogestrel - 91-day Levonorgestrel)

8. Secondary Outcome: Change From Baseline to End of Month 6 in Tissue Plasminogen Activator (t-PA)
Description: Tissue plasminogen activator catalyzes the conversion of plasminogen to plasmin, the major enzyme responsible for the breakdown of blood clots.
Time Frame: Baseline to Month 6
Population: Per-protocol population
Measure: Least Squares Mean (Standard Error); unit: µg/L
Arm/Group | 91-day Levonorgestrel Oral Contraceptive | 28-day Levonorgestrel Oral Contraceptive | 28-day Desogestrel Oral Contraceptive
Number analyzed (Participants) | 61 | 67 | 59
µg/L | -0.91 (0.32) | -1.48 (0.30) | -9.3 (0.32)
Statistical Analysis 1: Comparison: 91-day Levonorgestrel Oral Contraceptive vs 28-day Levonorgestrel Oral Contraceptive; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.194, Mixed Models Analysis; Treatment Difference = -0.57, 95% CI 2-sided [-1.4 to 0.3] — Treatment difference is calculated as (28-day Levonorgestrel - 91-day Levonorgestrel)
Statistical Analysis 2: Comparison: 91-day Levonorgestrel Oral Contraceptive vs 28-day Desogestrel Oral Contraceptive; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.967, Mixed Models Analysis; Treatment Difference = -0.02, 95% CI 2-sided [-0.9 to 0.9] — Treatment difference is calculated as (28-day Desogestrel - 91-day Levonorgestrel)

9. Secondary Outcome: Change From Baseline to End of Month 6 in Factor II
Description: Clotting factor II, also called prothrombin, functions in blood coagulation. Results are reported as percent of normal plasma concentrations. By definition, normal plasma contains 100% (1 unit/mL) of each factor. The reference range is approximately 60% to 140% for adults.
Time Frame: Baseline to Month 6
Population: Per-protocol population
Measure: Least Squares Mean (Standard Error); unit: percentage of normal
Arm/Group | 91-day Levonorgestrel Oral Contraceptive | 28-day Levonorgestrel Oral Contraceptive | 28-day Desogestrel Oral Contraceptive
Number analyzed (Participants) | 61 | 67 | 59
percentage of normal | 6.89 (1.73) | 7.98 (1.65) | 8.57 (1.76)
Statistical Analysis 1: Comparison: 91-day Levonorgestrel Oral Contraceptive vs 28-day Levonorgestrel Oral Contraceptive; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.648, Mixed Models Analysis; Treatment Difference = 1.09, 95% CI 2-sided [-3.6 to 5.8] — Treatment difference is calculated as (28-day Levonorgestrel - 91-day Levonorgestrel)
Statistical Analysis 2: Comparison: 91-day Levonorgestrel Oral Contraceptive vs 28-day Desogestrel Oral Contraceptive; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.496, Mixed Models Analysis; Treatment Difference = 1.68, 95% CI 2-sided [-3.2 to 6.6] — Treatment difference is calculated as (28-day Desogestrel - 91-day Levonorgestrel)

10. Secondary Outcome: Change From Baseline to End of Month 6 in Factor VII
Description: Clotting factor VII, also called proconvertin or autoprothrombin I, functions in blood coagulation.
  Results are reported as percent of normal plasma concentrations. By definition, normal plasma contains 100% (1 unit/mL) of each factor. The reference range is approximately 60% to 140% for adults.
Time Frame: Baseline to Month 6
Population: Per-protocol population
Measure: Least Squares Mean (Standard Error); unit: percentage of normal
Arm/Group | 91-day Levonorgestrel Oral Contraceptive | 28-day Levonorgestrel Oral Contraceptive | 28-day Desogestrel Oral Contraceptive
Number analyzed (Participants) | 61 | 67 | 59
percentage of normal | 14.27 (7.52) | 22.98 (7.18) | 43.22 (7.67)
Statistical Analysis 1: Comparison: 91-day Levonorgestrel Oral Contraceptive vs 28-day Levonorgestrel Oral Contraceptive; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.405, Mixed Models Analysis; Treatment Difference = 8.71, 95% CI 2-sided [-11.9 to 29.3] — Treatment difference is calculated as (28-day Levonorgestrel - 91-day Levonorgestrel)
Statistical Analysis 2: Comparison: 91-day Levonorgestrel Oral Contraceptive vs 28-day Desogestrel Oral Contraceptive; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.008, Mixed Models Analysis; Treatment Difference = 28.95, 95% CI 2-sided [7.7 to 50.2] — Treatment difference is calculated as (28-day Desogestrel - 91-day Levonorgestrel)

11. Secondary Outcome: Change From Baseline to End of Month 6 in Factor VIII
Description: Clotting factor VIII, also known as anti-hemophilic factor (AHF), functions in blood coagulation by stabilizing fibrin clots.
  Results are reported as a percent of the amount expected in normal plasma. By definition, the mean value in normal plasma is 100%. The reference range is approximately 70% to 140%.for adults.
Time Frame: Baseline to Month 6
Population: Per-protocol population
Measure: Least Squares Mean (Standard Error); unit: percentage of normal
Arm/Group | 91-day Levonorgestrel Oral Contraceptive | 28-day Levonorgestrel Oral Contraceptive | 28-day Desogestrel Oral Contraceptive
Number analyzed (Participants) | 61 | 67 | 59
percentage of normal | -3.23 (2.98) | 0.08 (2.87) | 5.53 (3.05)
Statistical Analysis 1: Comparison: 91-day Levonorgestrel Oral Contraceptive vs 28-day Levonorgestrel Oral Contraceptive; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.425, Mixed Models Analysis; Treatment Difference = 3.30, 195% CI 2-sided [-4.9 to 11.5] — Treatment difference is calculated as (28-day Levonorgestrel - 91-day Levonorgestrel)
Statistical Analysis 2: Comparison: 91-day Levonorgestrel Oral Contraceptive vs 28-day Desogestrel Oral Contraceptive; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.041, Mixed Models Analysis; Treatment Difference = 8.76, 95% CI 2-sided [0.3 to 17.2] — Treatment difference is calculated as (28-day Desogestrel - 91-day Levonorgestrel)

12. Secondary Outcome: Change From Baseline to End of Month 6 in Antithrombin
Description: Antithrombin is a protein in the blood that naturally blocks blood clots from forming.
  Results are reported as a percent of the amount expected in normal plasma. By definition, the mean value in normal plasma is 100%. The reference range is approximately 80% to 130%.for adults.
Time Frame: Baseline to Month 6
Population: Per-protocol population
Measure: Least Squares Mean (Standard Error); unit: percentage of normal
Arm/Group | 91-day Levonorgestrel Oral Contraceptive | 28-day Levonorgestrel Oral Contraceptive | 28-day Desogestrel Oral Contraceptive
Number analyzed (Participants) | 61 | 67 | 59
percentage of normal | 2.36 (1.00) | -0.05 (0.98) | -0.83 (1.03)
Statistical Analysis 1: Comparison: 91-day Levonorgestrel Oral Contraceptive vs 28-day Levonorgestrel Oral Contraceptive; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.088, Mixed Models Analysis; Treatment Difference = -2.40, 95% CI 2-sided [-5.2 to 0.4] — Treatment difference is calculated as (28-day Levonorgestrel - 91-day Levonorgestrel)
Statistical Analysis 2: Comparison: 91-day Levonorgestrel Oral Contraceptive vs 28-day Desogestrel Oral Contraceptive; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.028, Mixed Models Analysis; Treatment Difference = -3.19, 95% CI 2-sided [-6.0 to -0.3] — Treatment difference is calculated as (28-day Desogestrel - 91-day Levonorgestrel)

13. Secondary Outcome: Change From Baseline to End of Month 6 in Protein C Activity
Description: Protein C helps to regulate blood clot formation. Activated Protein C (APC) combines with Protein S (a cofactor) to degrade coagulation factors VIIIa and Va, slowing down the generation of new thrombin and inhibiting further clotting.
  Results are reported as a percent of the amount expected in normal plasma. By definition, the mean value in normal plasma is 100%. The reference range is approximately 70% to 140% for adults.
Time Frame: Baseline to Month 6
Population: Per-protocol population
Measure: Least Squares Mean (Standard Error); unit: percentage of normal
Arm/Group | 91-day Levonorgestrel Oral Contraceptive | 28-day Levonorgestrel Oral Contraceptive | 28-day Desogestrel Oral Contraceptive
Number analyzed (Participants) | 61 | 67 | 59
percentage of normal | -6.15 (2.62) | -4.39 (2.53) | -2.41 (2.70)
Statistical Analysis 1: Comparison: 91-day Levonorgestrel Oral Contraceptive vs 28-day Levonorgestrel Oral Contraceptive; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.631, Mixed Models Analysis; Treatment Difference = 1.75, 95% CI 2-sided [-5.4 to 8.9] — Treatment difference is calculated as (28-day Levonorgestrel - 91-day Levonorgestrel)
Statistical Analysis 2: Comparison: 91-day Levonorgestrel Oral Contraceptive vs 28-day Desogestrel Oral Contraceptive; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.323, Mixed Models Analysis; Treatment Difference = 3.73, 95% CI 2-sided [-3.7 to 11.2] — Treatment difference is calculated as (28-day Desogestrel - 91-day Levonorgestrel)

14. Secondary Outcome: Change From Baseline to End of Month 6 in Protein C Antigen
Description: Protein C helps to regulate blood clot formation. Activated Protein C (APC) combines with Protein S (a cofactor) to degrade coagulation factors VIIIa and Va, slowing down the generation of new thrombin and inhibiting further clotting.
  Results are reported as a percent of the amount expected in normal plasma. By definition, the mean value in normal plasma is 100%. The reference range is approximately 70% to 140% in adults.
Time Frame: Baseline to Month 6
Population: Per-protocol population
Measure: Least Squares Mean (Standard Error); unit: percentage of normal
Arm/Group | 91-day Levonorgestrel Oral Contraceptive | 28-day Levonorgestrel Oral Contraceptive | 28-day Desogestrel Oral Contraceptive
Number analyzed (Participants) | 61 | 67 | 59
percentage of normal | 12.83 (2.26) | 11.97 (2.17) | 10.00 (2.32)
Statistical Analysis 1: Comparison: 91-day Levonorgestrel Oral Contraceptive vs 28-day Levonorgestrel Oral Contraceptive; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.783, Mixed Models Analysis; Treatment Difference = -0.86, 595% CI 2-sided [-7.0 to 5.3] — Treatment difference is calculated as (28-day Levonorgestrel - 91-day Levonorgestrel)
Statistical Analysis 2: Comparison: 91-day Levonorgestrel Oral Contraceptive vs 28-day Desogestrel Oral Contraceptive; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.384, Mixed Models Analysis; Treatment Difference = -2.83, 95% CI 2-sided [-9.2 to 3.6] — Treatment difference is calculated as (28-day Desogestrel - 91-day Levonorgestrel)

15. Secondary Outcome: Change From Baseline to End of Month 6 in Free Protein S
Description: Protein S helps to regulate blood clot formation. Protein S exists in two forms: a free form and a complex form. Free protein S combines with Protein C to degrade coagulation factors VIIIa and Va, slowing down the generation of new thrombin and inhibiting further clotting.
  Results are reported as a percent of the amount expected in normal plasma. By definition, the mean value in normal plasma is 100%. The reference range is approximately 70% to 140%; lower for women than for men.
Time Frame: Baseline to Month 6
Population: Per-protocol population
Measure: Least Squares Mean (Standard Error); unit: percentage of normal
Arm/Group | 91-day Levonorgestrel Oral Contraceptive | 28-day Levonorgestrel Oral Contraceptive | 28-day Desogestrel Oral Contraceptive
Number analyzed (Participants) | 61 | 67 | 59
percentage of normal | 2.96 (2.13) | 4.62 (2.03) | -18.2 (2.17)
Statistical Analysis 1: Comparison: 91-day Levonorgestrel Oral Contraceptive vs 28-day Levonorgestrel Oral Contraceptive; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.572, Mixed Models Analysis; Treatment Difference = 1.66, 95% CI 2-sided [-4.1 to 7.5] — Treatment difference is calculated as (28-day Levonorgestrel - 91-day Levonorgestrel)
Statistical Analysis 2: Comparison: 91-day Levonorgestrel Oral Contraceptive vs 28-day Desogestrel Oral Contraceptive; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Treatment Difference = -20.98, 95% CI 2-sided [-27.0 to -15.0] — Treatment difference is calculated as (28-day Desogestrel - 91-day Levonorgestrel)

16. Secondary Outcome: Change From Baseline to End of Month 6 in Total Protein S
Description: Protein S helps to regulate blood clot formation. Protein S exists in two forms: a free form and a complex form. Free protein S combines with activated protein C to degrade coagulation factors VIIIa and Va, slowing down the generation of new thrombin and inhibiting further clotting.
  Results are reported as a percent of the amount expected in normal plasma. By definition, the mean value in normal plasma is 100%. The reference range is approximately 70% to 140%; lower for women than for men.
Time Frame: Baseline to Month 6
Population: Per-protocol population
Measure: Least Squares Mean (Standard Error); unit: percentage of normal
Arm/Group | 91-day Levonorgestrel Oral Contraceptive | 28-day Levonorgestrel Oral Contraceptive | 28-day Desogestrel Oral Contraceptive
Number analyzed (Participants) | 61 | 67 | 59
percentage of normal | -11.06 (1.51) | -11.48 (1.45) | -21.59 (1.55)
Statistical Analysis 1: Comparison: 91-day Levonorgestrel Oral Contraceptive vs 28-day Levonorgestrel Oral Contraceptive; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.841, Mixed Models Analysis; Treatment Difference = -0.42, 95% CI 2-sided [-4.6 to 3.7] — Treatment difference is calculated as (28-day Levonorgestrel - 91-day Levonorgestrel)
Statistical Analysis 2: Comparison: 91-day Levonorgestrel Oral Contraceptive vs 28-day Desogestrel Oral Contraceptive; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Treatment Difference = -10.53, 95% CI 2-sided [-14.8 to -6.3] — Treatment difference is calculated as (28-day Desogestrel - 91-day Levonorgestrel)

17. Secondary Outcome: Change From Baseline to End of Month 6 in Tissue Factor Pathway Inhibitor (TFPI)
Description: Tissue Factor Pathway Inhibitor (TFPI) is an anti-coagulation protein that binds to activated protein X.
Time Frame: Baseline to Month 6
Population: Per-protocol population
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | 91-day Levonorgestrel Oral Contraceptive | 28-day Levonorgestrel Oral Contraceptive | 28-day Desogestrel Oral Contraceptive
Number analyzed (Participants) | 61 | 67 | 59
ng/mL | 4.65 (1.26) | 2.54 (1.21) | -1.34 (1.30)
Statistical Analysis 1: Comparison: 91-day Levonorgestrel Oral Contraceptive vs 28-day Levonorgestrel Oral Contraceptive; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.227, Mixed Models Analysis; Treatment Difference = -2.11, 95% CI 2-sided [-5.6 to 1.3] — Treatment difference is calculated as (28-day Levonorgestrel - 91-day Levonorgestrel)
Statistical Analysis 2: Comparison: 91-day Levonorgestrel Oral Contraceptive vs 28-day Desogestrel Oral Contraceptive; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis; Treatment Difference = -5.99, 95% CI 2-sided [-9.6 to -2.4] — Treatment difference is calculated as (28-day Desogestrel - 91-day Levonorgestrel)

18. Secondary Outcome: Change From Baseline to End of Month 6 in Thyroid Stimulating Hormone (TSH)
Time Frame: Baseline top Month 6
Population: Per-protocol population with available data
Measure: Least Squares Mean (Standard Error); unit: mIU/L
Arm/Group | 91-day Levonorgestrel Oral Contraceptive | 28-day Levonorgestrel Oral Contraceptive | 28-day Desogestrel Oral Contraceptive
Number analyzed (Participants) | 61 | 67 | 58
mIU/L | -0.22 (0.13) | 0.10 (0.13) | 0.22 (0.13)
Statistical Analysis 1: Comparison: 91-day Levonorgestrel Oral Contraceptive vs 28-day Levonorgestrel Oral Contraceptive; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.076, Mixed Models Analysis; Treatment Difference = 0.33, 95% CI 2-sided [-0.0 to 0.7] — Treatment difference is calculated as (28-day Levonorgestrel - 91-day Levonorgestrel)
Statistical Analysis 2: Comparison: 91-day Levonorgestrel Oral Contraceptive vs 28-day Desogestrel Oral Contraceptive; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.021, Mixed Models Analysis; Treatment Difference = 0.44, 95% CI 2-sided [0.1 to 0.8] — Treatment difference is calculated as (28-day Desogestrel - 91-day Levonorgestrel)

19. Secondary Outcome: Change From Baseline to End of Month 6 in Total Cortisol
Time Frame: Baseline to Month 6
Population: Per-protocol population
Measure: Least Squares Mean (Standard Error); unit: nmol/L
Arm/Group | 91-day Levonorgestrel Oral Contraceptive | 28-day Levonorgestrel Oral Contraceptive | 28-day Desogestrel Oral Contraceptive
Number analyzed (Participants) | 61 | 67 | 59
nmol/L | 217.94 (24.39) | 262.40 (23.39) | 227.68 (24.96)
Statistical Analysis 1: Comparison: 91-day Levonorgestrel Oral Contraceptive vs 28-day Levonorgestrel Oral Contraceptive; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.190, Mixed Models Analysis; Treatment Difference = 44.46, 95% CI 2-sided [-22.3 to 111.2] — Treatment difference is calculated as (28-day Levonorgestrel - 91-day Levonorgestrel)
Statistical Analysis 2: Comparison: 91-day Levonorgestrel Oral Contraceptive vs 28-day Desogestrel Oral Contraceptive; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.781, Mixed Models Analysis; Treatment Difference = 9.74, 95% CI 2-sided [-59.4 to 78.9] — Treatment difference is calculated as (28-day Desogestrel - 91-day Levonorgestrel)

20. Secondary Outcome: Change From Baseline to End of Month 6 in Corticosteroid Binding Globulin
Time Frame: Baseline to Month 6
Population: Per-protocol population with available data
Measure: Least Squares Mean (Standard Error); unit: nmol/L
Arm/Group | 91-day Levonorgestrel Oral Contraceptive | 28-day Levonorgestrel Oral Contraceptive | 28-day Desogestrel Oral Contraceptive
Number analyzed (Participants) | 61 | 67 | 58
nmol/L | 576.33 (45.37) | 563.85 (43.41) | 634.64 (46.74)
Statistical Analysis 1: Comparison: 91-day Levonorgestrel Oral Contraceptive vs 28-day Levonorgestrel Oral Contraceptive; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.843, Mixed Models Analysis; Treatment Difference = -12.49, 95% CI 2-sided [-136.4 to 111.4] — Treatment difference is calculated as (28-day Levonorgestrel - 91-day Levonorgestrel)
Statistical Analysis 2: Comparison: 91-day Levonorgestrel Oral Contraceptive vs 28-day Desogestrel Oral Contraceptive; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.376, Mixed Models Analysis; Treatment Difference = 58.30, 95% CI 2-sided [-71.3 to 187.9] — Treatment difference is calculated as (28-day Desogestrel - 91-day Levonorgestrel)

21. Secondary Outcome: Change From Baseline to End of Month 6 in Sex Hormone Binding Globulin (SHBG)
Time Frame: Baseline to Month 6
Population: Per-protocol population with available data
Measure: Least Squares Mean (Standard Error); unit: mIU/L
Arm/Group | 91-day Levonorgestrel Oral Contraceptive | 28-day Levonorgestrel Oral Contraceptive | 28-day Desogestrel Oral Contraceptive
Number analyzed (Participants) | 61 | 66 | 58
mIU/L | 34.87 (8.40) | 30.85 (8.08) | 165.01 (8.67)
Statistical Analysis 1: Comparison: 91-day Levonorgestrel Oral Contraceptive vs 28-day Levonorgestrel Oral Contraceptive; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.731, Mixed Models Analysis; Treatment Difference = -4.01, 95% CI 2-sided [-27.0 to 19.0] — Treatment difference is calculated as (28-day Levonorgestrel - 91-day Levonorgestrel)
Statistical Analysis 2: Comparison: 91-day Levonorgestrel Oral Contraceptive vs 28-day Desogestrel Oral Contraceptive; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Treatment Difference = 130.15, 95% CI 2-sided [106.2 to 154.1] — Treatment difference is calculated as (28-day Desogestrel - 91-day Levonorgestrel)

ADVERSE EVENTS:
Time Frame: From the first dose of study drug until 14 days after the last dose (up to 27 weeks).
Arm/Group | 91-day Levonorgestrel Oral Contraceptive | 28-day Levonorgestrel Oral Contraceptive | 28-day Desogestrel Oral Contraceptive
Serious Adverse Events (participants affected / at risk) | 0/83 | 0/89 | 0/80
Other Adverse Events (participants affected / at risk) | 16/83 | 10/89 | 17/80
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 91-day Levonorgestrel Oral Contraceptive (N=83) | 28-day Levonorgestrel Oral Contraceptive (N=89) | 28-day Desogestrel Oral Contraceptive (N=80)
Nausea (Gastrointestinal disorders) | 5 (5) | 4 (5) | 8 (9)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 4 (4)
Prothrombin level increased (Investigations) | 0 (0) | 1 (1) | 4 (4)
Headache (Nervous system disorders) | 3 (3) | 1 (1) | 4 (4)
Metrorrhagia (Reproductive system and breast disorders) | 11 (14) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.